## The University of New Mexico Health Sciences Center Consent and Authorization to Participate in a Research Study Effects of the COVID-19 Health Emergency on the Biopsychosocial Health of Rural Residents of New Mexico using Mixed Methods

## Dear Prospective Participant,

Researchers at the University of New Mexico are inviting you to take part in a quality of life survey and interview/questionnaire about your perceptions of the COVID-19 health emergency. We want to understand how the health emergency is affecting you and your family. We are attempting to reach a representative sample of New Mexico residents across rural and urban New Mexico, and that is why you are being asked to participate in this research. The name of this project is: Effects of the COVID-19 Health Emergency on the Biopsychosocial Health of Rural Residents of New Mexico using Mixed Methods.

## WHAT ARE THE KEY REASONS YOU MIGHT CHOOSE TO VOLUNTEER FOR THIS STUDY?

Although you may not get personal benefit from taking part in this research study, your responses may help us understand more about how people are coping with the COVID-19 health emergency. This knowledge may help health care organizations and government institutions improve services and assistance to people in the future.

## WHAT ARE THE KEY REASONS YOU MIGHT NOT CHOOSE TO VOLUNTEER FOR THIS STUDY?

Reasons to choose NOT to volunteer for the study may include not wanting to be asked questions that make you feel uncomfortable or cause you to become upset or that you do not feel you have the time to participate in the study.

The quality of life survey will take about 10-12 minutes to complete. The interview/questionnaire will take from about 30 minutes to 1 hour.

There are no known risks to participating in this study. Although we have tried to minimize this, some questions may make you upset or feel uncomfortable and you may choose not to answer them. If some questions do upset you, we can tell you about some people who may be able to help you with these feelings.

Your response to the survey and interview/questionnaire is anonymous which means no names will appear or be used on research documents or be used in presentations or publications. The research team will not know that any information you provided came from you, nor even whether you participated in the study. Your responses to the survey will be kept confidential to the extent allowed by law. Study records will be maintained for 3 years after the study closes. When we write about the study and its results you will not be identified.

We hope to receive completed questionnaires from about 300 people living in New Mexico, so your answers are important to us. Of course, you have a choice about whether or not to complete the survey/questionnaire, but if you do participate, you are free to skip any questions or discontinue at any time.

If you have questions about the study, please feel free to ask; my contact information is given below. If you have questions regarding your legal rights as a research subject, you may call the UNM Human Research Protections Office at (505) 272-1129.

HRRC# 20-266 Version date: 05/05/2020

Thank you in advance for your assistance with this important project. If you could complete the survey and questionnaire and return within seven days, it will be very appreciated. To ensure your responses/opinions will be included, please use the enclosed postage paid envelope to return your completed survey/questionnaire. By returning this survey by mail **OR** by talking to us by phone, you will be agreeing to participate in the above described research study.

Sincerely,

Carla Wilhite, OTD, OTR/L
Assistant Professor
Department of Pediatrics-Occupational Therapy Graduate Program
University of New Mexico Health Sciences
PHONE: 505-272-3324

E-MAIL: cwilhite@salud.unm.edu

HRRC# 20-266 Version date: 05/05/2020